CLINICAL TRIAL: NCT01073267
Title: A Phase II Study of Total Skin Electron Beam Therapy (TSEBT) to Dose of 12 Gy in Stage IB-IIIA Mycosis Fungoides
Brief Title: Study of Total Skin Electron Beam Therapy (TSEBT) in Stage IB-IIIA Mycosis Fungoides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0444; NCI-2011-00560 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma
Keywords: Stage IB-IIIA Mycosis fungoides; Total Skin Electron Beam Therapy; TSEBT
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TSEBT (Experimental): Total Skin Electron Beam Therapy (TSEBT) to dose of 12 Gy
  Interventions: Radiation: TSEBT

INTERVENTIONS:
Radiation: TSEBT — Total skin electron beam therapy (TSEBT) to a total dose of 12 Gray (TSEBT 12 Gy), low-dose radiation to the skin 4-5 days a week for 3 weeks.

SUMMARY:
The goal of this clinical research study is to learn if a lower than standard dose of total skin electron beam radiation therapy to the skin can help to control mycosis fungoides. The safety of this dose level will also be studied.

DETAILED DESCRIPTION:
Study Radiation:

During total skin electron beam therapy, radiation is given to the entire surface of the skin. This may cause the cancer cells to die.

Researchers would like to learn the level of effectiveness of this lower dose of radiation therapy because it is likely to have fewer side effects than the standard, higher dose.

Screening Period:

Signing this consent form does not mean that you will be able to take part in this study. You will have the following "screening tests" to help the doctor decide if you are eligible to take part in this study.

Within 6 weeks before the radiation therapy can begin:

* If the doctor thinks it is needed, you will have a computed tomography (CT) scan or other type of scan to check the status of the disease.
* If the doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to check for cancer in your lymph nodes.

Within 4 weeks before the radiation therapy can begin:

* Your medical history will be recorded, including any drugs you are taking and have taken.
* You will have a physical exam, including a skin exam and measurement of your weight and vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will be asked how well you are able to perform the normal activities of daily living (performance status).
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Women who are able to become pregnant must have a negative urine pregnancy test.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Wash-Out Period:

If you agree to take part in this study, from that day until your first study radiation treatment, you will stop certain treatments for mycosis fungoides. This is called a "wash-out period". The number of weeks will be different depending on what treatments you may be receiving. The study doctor will explain the types of treatments and schedule for stopping them.

* For the 2 weeks before radiation, you will stop using any cancer drugs that are "topical" (applied onto the skin).
* For the 4 weeks before radiation, you will stop any radiation therapy, phototherapy (cancer treatments with light), cancer drugs that are "systemic" (affecting the whole body), and any other investigational therapy.

Study Visit Before Radiation Therapy:

Within 1 week before your first radiation treatment, the following tests and procedures will be performed:

-You will have a physical exam, including a skin exam and measurement of your weight and vital signs.

Your performance status will be recorded.

* You will be asked about any drugs you may be taking.
* The doctor will draw on your skin with a marker to mark areas of your body that are unexposed. This is to help plan the radiation treatments. Depending on your body shape, about 8-16 body areas will be marked.
* Photos will be taken of your whole body. These photos will be used to help the doctor find out how much skin is affected by the disease.

Radiation Treatments:

If you are found to be eligible to take part in this study, you will receive low-dose radiation to the skin 4-5 days a week for 3 weeks.

On Mondays and Tuesdays, you will receive radiation that can cover your entire skin area. You will be standing during the treatment. This wider-field radiation treatment cannot give enough radiation to the unexposed areas of your body, such as under the arms, under the breasts for females, under the belly, in the private areas, and the soles of the feet. For this reason, in addition to the wider-field radiation, you will also receive radiation that covers these smaller areas of your body on Wednesdays and Thursdays. The amount of radiation that these smaller body areas will receive is designed to be the same as the amount the rest of the skin will receive.

If the study doctor thinks it is needed for standard care, you will also receive radiation treatments on other tumors. In most cases, this will be on Fridays. It will be 4-7 treatments, depending on the tumor size.

At Weeks 2 and 3 of radiation treatment, you will be asked about any side effects that have occurred.

Length of Study:

You may receive up to 3 weeks of low-dose radiation therapy. You will be taken off the study treatment early if intolerable side effects occur or the disease gets worse. The follow-up period in this study lasts up to 12 months after the last treatment.

Follow-Up and End-of-Study Visits:

After your last dose of low-dose radiation therapy, you will have follow-up visits 1 to 3 weeks after treatment, every 2 months for 6 months, and then every 3 months for a total of 12 months. However, if the disease gets worse during this 12-month follow-up period, the follow-up visits will stop. When you are off-study, an end-of-study visit will occur.

If you stopped the radiation early due to intolerable side effects, you will have follow-up visits twice a week until the doctor thinks the side effects have gotten better. After that, you will return for an end-of-study visit.

At the follow-up visits and end-of-study visit, the following tests and procedures will be performed:

* You will have a physical exam, including a skin exam and measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and side effects that may have occurred.
* Photos will be taken of your whole body to check the status of the disease.
* Blood (about 1 teaspoon) will be drawn for routine tests

This is an investigational study. For this type of cancer, the dose of radiation in this study is lower than standard. The type of radiation therapy (total skin electron beam therapy) is standard. At this time, the lower dose is only being used in research.

Up to 20 patients will be take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed mycosis fungoides in stage IB-IIIA
2. Patients must have failed or have been intolerant to at least one prior systemic or topical therapy which may include topical steroids
3. 18 years of age or older
4. Life expectancy greater than 6 months
5. Eastern Cooperative Oncology Group (ECOG) of </= 2
6. Adequate bone marrow function: White blood count (WBC) >/= 2000/uL; platelet count>/= 100,000/mm3; Absolute neutrophil count (ANC) >/= 1000
7. Required wash out period for prior therapies (Note: patients with progressive disease may be treated earlier than required washout period per Investigator's decision) a) Topical therapy: 2 weeks, b) Systemic biologic, monoclonal antibody or chemotherapy: 4 weeks, c) Radiotherapy (excluding TSEBT) or phototherapy: 4 weeks, d) Other investigational therapy: 4 weeks
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior courses of TSEBT (Note: localized skin-directed radiotherapy is allowed if administered at least 4 weeks prior to initiation on study)
2. Underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of patient to undergo treatment
3. Prior malignancy (active within 5 years of screening) except completely excised non-invasive basal cell or squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix
4. Pregnant or lactating
5. Initiation or change in dosage of topical corticosteroids within 3 weeks of study treatment (Note: topical steroid use within 3 weeks is allowed provided the strength and use has been stable for at least 1 month; 'prescription strength' topical corticosteroids cannot be started during the study)
6. Any other medical history, including laboratory results, deemed by the Investigator to be likely to interfere with patient participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina Dabaja, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: February 19, 2010 to April 19, 2011. All participants recruited at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | TSEBT
Started | 4
Completed | 1
Not Completed | 3
Not completed — Disease Progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | TSEBT
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 69 [48 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate defined as the proportion of participants achieving complete clinical response (CCR) and partial response (PR) (i.e. overall response (OR)) as assessed by the modified Severity-Weighted Assessment Tool (mSWAT).
  Clinical response (according to mSWAT) are documented as stable disease (SD), partial response (PR), complete clinical response (CCR), or progressive disease (PD) as defined: Complete clinical response (CCR): no evidence of cutaneous disease on exam, confirmed at 4 week time point; Partial response (PR): ≥ 50% decrease of modified SWAT score compared to baseline score, confirmed at 4 week time point; Stable disease (SD): Neither CR, PR, or PD, i.e. change from baseline is less than 50% decrease, but also less than 25% increase in mSWAT score compared to nadir score; Progressive disease (PD): ≥ 25% increase in modified SWAT score compared with nadir score.
Time Frame: Baseline and at least 2 months
Population: Intent to treat population.
Measure: Number; unit: proportion of participants
Arm/Group | TSEBT
Number analyzed (Participants) | 4
proportion of participants | .25

ADVERSE EVENTS:
Time Frame: Adverse event information collected during the 3-week treatment period and for 3 months following completion of TSEBT (this applies to participants who withdraw from the study).
Arm/Group | TSEBT
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSEBT (N=4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Dermatology/Skin (Other (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Vision blurred (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Ocular/Visual (Other) (Eye disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Fat atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes